CLINICAL TRIAL: NCT05160519
Title: Class IV Laser Therapy on Ejection Fraction, Cardio Biomarkers and Functional Outcomes Among Individuals With Acute Coronary Syndrome
Brief Title: Class IV Laser Therapy on Ejection Fraction, Cardio Biomarkers and Functional Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asir John Samuel (Other)
Collaborators: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMDU/IEC/2157; U1111-1270-8393 (Other: Universal Trial Number (UTN)-WHO)
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Class IV Laser; ACS; Ejection fraction; Cardiac Biomarkers
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 30 participants will be irradiated with Class IV laser therapy over the left parasternal area to examine the effectiveness of Class IV laser.
  Interventions: Radiation: Class IV Laser
- Sham Controlled (Sham Comparator): 30 participants will subject to irradiation but the equipment will be kept off.
  Interventions: Radiation: Sham Class IV Laser

INTERVENTIONS:
Radiation: Class IV Laser — 30 participants will be irradiated with Class IV laser therapy over the left parasternal area to examine the efficacy of class IV laser on ejection fraction, Cardiac Biomarker and functional outcomes.
  Device: Litecure LCT-1000C Class IV laser will be used in contact method over the left parasternal area in 2nd, 3rd intercostal space and apex. Dosage and Parameters for the irradiation will be calculated. Parameters: 1. Wavelength: 980nm, 2. Power/ Energy density: 6W/6J/cm2 3. Frequency: CW 4. Energy delivered at each spot: 360J 5. irradiation spots: 3 6. Irradiation time: 60 sec at each spot.
  Both the patient and laser giver will use the laser protected eye wears to ensure standard practice for the laser.
  Arms: Experimental
Radiation: Sham Class IV Laser — 30 participants in sham control group will be suppose to irradiate with Class IV laser therapy over the left parasternal area, but the radiation will not be delivered.
  Device: Litecure LCT-1000C Class IV laser will be placed over the left parasternal area in 2nd, 3rd intercostal space and apex without switching on the instrument.
  Both the patient and laser giver will use the laser protected eye wears to ensure standard practice for the laser.
  Arms: Sham Controlled

SUMMARY:
A total of 60 Individuals with Acute coronary Syndrome who underwent angioplasty with or without stent will be recruited by purposive sampling method in a randomized double-blinded sham controlled trial. Recruited participants will be divided into two group of equal size (n = 30): Sham control group and experimental group by block randomization. The experimental group will subject to Class IV laser therapy along with the standard treatment regime at three spot(s) over the pericardium (left parasternal 2nd, 3rd intercostal space and apex) for a duration of 60 seconds at each point.; immediately after the angioplasty and subsequent two days. Left ventricular ejection fraction will be assessed at base line and after 3 days post-interventions. Cardiac biomarker (Troponin I) will be assessed at base line, peak hours (at 10 hour after revascularization) and on third day post intervention. Function outcomes will be assessed at baseline and at one month follow up.

DETAILED DESCRIPTION:
Individuals with acute coronary syndrome admitted in the Cardiac Care Unit of MMIMSR, Mullana, Ambala, Haryana who underwent angioplasty with or without stent during the study period will be screened according to selection criteria. Then the invited participants will be asked to sign a written informed consent for voluntarily participation in the study. Participants will be divided into two group of equal size (n = 30): Sham control group and experimental group by block randomization. The researcher will be divided into therapist and evaluator or assessor. The therapist will responsible for conducting the therapy and evaluator or assessor will responsible for assessment of outcome measures both pre and post intervention. All the assessor or evaluator (lab technicians who assess cardiac biomarkers, Cardiologist who perform echocardiography and assess ECG) will be blinded from the grouping of the participants. The participants will also be blinded to the study by use of laser protected eye wears. Left ventricular ejection fraction, cardiac biomarker (Troponin I) and functional outcomes will be assessed at base line. The experimental group will subject to Class IV laser therapy along with the standard treatment regime at three spot(s) over the pericardium (left parasternal 2nd, 3rd intercostal space and apex) for a duration of 60 seconds at each point.; immediately after the angioplasty and subsequent two days. The sham group will subject to irradiation but the equipment will be kept off. All the outcomes measures will be reassess after 3 days post-interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with Acute Coronary Syndrome (ACS) who underwent angioplasty with drug eluting implant
2. Both male and female above 18 years of age,
3. Hemodynamically stable,
4. Who voluntarily signed the informed consent.

Exclusion Criteria:

1. Tumor or growth around mediastinum,
2. Temporary or permanent pacemaker,
3. Receiving steroids or photosensitive drugs,
4. Pregnancy,
5. Epilepsy,
6. LVEF ≤ 30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction | changes will be measured at baseline and on 3rd day post intervention
  Left Ventricular ejection fraction is a is a direct indicator of left ventricle systolic function.
Cardiac Biomarker | changes will be measured at baseline, peak hours (10 hours post revascularization) and on 3rd day post intervention
  Cardiac Biomarkers (Troponin I) are the early markers of acute myocardial injury
Functional outcomes | changes will be measured at baseline and on one month follow up
  Hindi version of Seattle angina Questionnaire will be used to assess functional outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep K Jangra, PhD Scholar, Principal Investigator — M.M. Institute of Physiotherapy & Rehabilitation, (Maharishi Markandeshwar Deemed to be University); Asir J Samuel, PhD, Study Director — M.M. Institute of Physiotherapy & Rehabilitation, (Maharishi Markandeshwar Deemed to be University); Anupam Bhambhani, DM, Study Director — MMIMSR, Maharishi Markandeshwar Deemed to be University
Locations (1):
- Mandeep Kumar Jangra, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liebert A, Krause A, Goonetilleke N, Bicknell B, Kiat H. A Role for Photobiomodulation in the Prevention of Myocardial Ischemic Reperfusion Injury: A Systematic Review and Potential Molecular Mechanisms. Sci Rep. 2017 Feb 9;7:42386. doi: 10.1038/srep42386. PMID 28181487
- [Background] Kazemi Khoo N, Babazadeh K, Lajevardi M, Dabaghian FH, Mostafavi E. Application of Low-Level Laser Therapy Following Coronary Artery Bypass Grafting (CABG) Surgery. J Lasers Med Sci. 2014 Spring;5(2):86-91. PMID 25653805
- [Background] Elbaz-Greener G, Sud M, Tzuman O, Leitman M, Vered Z, Ben-Dov N, Oron U, Blatt A. Adjunctive laser-stimulated stem-cells therapy to primary reperfusion in acute myocardial infarction in humans: Safety and feasibility study. J Interv Cardiol. 2018 Dec;31(6):711-716. doi: 10.1111/joic.12539. Epub 2018 Jul 12. PMID 29999208
- [Background] Quirk BJ, Sonowal P, Jazayeri MA, Baker JE, Whelan HT. Cardioprotection from ischemia-reperfusion injury by near-infrared light in rats. Photomed Laser Surg. 2014 Sep;32(9):505-11. doi: 10.1089/pho.2014.3743. Epub 2014 Aug 5. PMID 25093393